CLINICAL TRIAL: NCT00715039
Title: A 4-Week, Double-Blind, Randomized, Multicenter, Fixed Dose, Placebo-Controlled, Parallel Group Study of Lorazepam and Paroxetine in Patients With Generalized Anxiety Disorder: Assessment of a New Instrument Intended to Capture Rapid Onset
Brief Title: Clinical Study Assessing a New Scale to Measure Onset of Action in Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: A9001141
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-10

CONDITIONS: Anxiety Disorders
Keywords: generalized anxiety disorder; onset of efficacy; Daily Assessment of Symptoms-Anxiety (DAS-A); Methods
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Lorazepam; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- lorazepam (Active Comparator)
  Interventions: Drug: lorazepam
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- paroxetine (Active Comparator)
  Interventions: Drug: paroxetine

INTERVENTIONS:
Drug: lorazepam — 1.0 mg p.o. three times a day for three days, then 1.5mg p.o. three times a day for 25 days
  Other Names: Ativan
  Arms: lorazepam
Drug: placebo — placebo p.o. t.i.d. for 28 days; placebo matching lorazepam and paroxetine
  Arms: placebo
Drug: paroxetine — 20mg p.o. daily for 28 days; and matching placebo twice a day to maintain blind
  Other Names: Paxil
  Arms: paroxetine

SUMMARY:
The study is to assess the performance characteristics of a new measure to assess onset of efficacy in a GAD patient population.

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnosis of GAD (DSM IV, 300.02) as established by the clinician using all sources of data including the MINI structured interview
* HAM A score ³20 at the Screening (Study Day -7) and Baseline (Study Day 1) Visits by observer rating
* Good health as determined by medical history, physical examination, vital signs, electrocardiography (ECG), and clinical laboratory measurements
* Covi Anxiety Scale total score ³9 and Raskin Depression Scale total score £7 at the Screening Visit (to ensure predominance of anxiety symptoms over depression symptoms)
* Age 18 to 65 (inclusive)

Exclusion Criteria:

* Patients with most other current DSM-IV Axis I disorders.
* Patients with current or past schizophrenia, Psychotic disorder
* Delirium, dementia, amnestic, and other clinically significant cognitive disorders
* Bipolar or schizoaffective disorder
* Benzodiazepine abuse or dependence; and/or Factitious disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2003-10; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Average change from baseline over the first 6 days of treatment assessment (Study Days 2 through 7) on the Daily Assessment of Symptoms - Anxiety (DAS-A) questionnaire. | baseline, days 2 through 7

SECONDARY OUTCOMES:
CGIC at endpoint (LOCF) | endpoint
PGIC at endpoint (LOCF) | endpoint
Q-LES-Q change from baseline to endpoint (LOCF) | baseline, endpoint
SF-36v2 Mental Health change from baseline to endpoint (LOCF) | baseline, endpoint
HADS-A change from baseline to endpoint (LOCF) | baseline, endpoint
HADS-D change from baseline to endpoint (LOCF) | baseline, endpoint
Change from baseline to endpoint (Weeks 1, 2, 4, and 5) in the HAM-A total score. | baseline and weeks 1,2,4, and 5
Change from baseline to daily time point (Study Days 2 through 7) on the DAS-A. | baseline and days 2 through 7
DAS-A change from baseline to endpoint (LOCF) | baseline to endpoint
DAS-A 30% and 50% improvement at endpoint; | endpoint
DAS-A 30% sustained improvement beginning at week 1 | baseline, week1, 2,4,
HAM-A 30% sustained improvement beginning at week 1 | baseline, weeks 1,2,4
HAM-A 30% and 50% improvement at endpoint | endpoint
GA-VAS average change from baseline over the first 6 days | baseline, days 2-7
Change from baseline to daily time point on the GA-VAS(study days 2 through 7) | baseline, days 2-7
GA-VAS change from baseline to endpoint | aseline, endpoint
GA-VAS sustained 30% improvement beginning at week 1 | baseline, weeks 1,2,4
GA-VAS 30% and 50% improvement at endpoint | endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Sherman Oaks, California
  - Pfizer Investigational Site, Van Nuys, California
  - Pfizer Investigational Site, Casselberry, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Cincinnati, Ohio

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001141&StudyName=Clinical%20study%20assessing%20a%20new%20scale%20to%20measure%20onset%20of%20action%20in%20Generalized%20Anxiety%20Disorder